CLINICAL TRIAL: NCT04736394
Title: A Multi-center, Randomized, Open-label, Parallel-controlled Phase 3 Clinical Trial to Evaluate the Clinical Safety and Efficacy of APL-1202 as a Single-agent Oral Treatment Versus Intravesical Instillation of Epirubicin Hydrochloride in naïve Intermediate-risk Non-muscle Invasive Bladder Cancer (NMIBC) Patients
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of APL-1202 as a Single-agent Oral Treatment Versus Intravesical Instillation of Epirubicin Hydrochloride in naïve Intermediate-risk NMIBC Patients
Acronym: ASCERTAIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YHCT-NIT-R2
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epirubicin hydrochloride group (Active Comparator): intravesical instillation of Epirubicin hydrochloride
  Interventions: Drug: Epirubicin Hydrochloride
- APL-1202 group (Experimental): receive APL-1202 single-agent oral treatment
  Interventions: Drug: APL-1202

INTERVENTIONS:
Drug: APL-1202 — APL-1202 single-agent oral treatment
  Arms: APL-1202 group
Drug: Epirubicin Hydrochloride — Epirubicin hydrochloride
  Arms: Epirubicin hydrochloride group

SUMMARY:
A multi-center, randomized, open-label, parallel-controlled Phase Ⅲ clinical trial to evaluate the clinical safety and efficacy of APL-1202 as a single-agent oral treatment versus intravesical instillation of Epirubicin hydrochloride in naïve intermediate-risk non-muscle invasive bladder cancer (NMIBC) patients

DETAILED DESCRIPTION:
A multi-center, randomized, open-label, placebo controlled Phase Ⅲ trial. The subjects must be histopathologically diagnosed, naïve intermediate-risk NMIBC patient. The screening period is 6 weeks prior to treatment.

The trial including 2 stages:

• First stages: The subjects are randomly assigned to receive APL-1202 single-agent oral treatment or intravesical instillation of Epirubicin hydrochloride at a ratio of 1:1. At this stage, an interim analysis will be performed after the first 100 subjects enrolled completing the 6-month visit (completing the second cystoscopy), and the Independent Data Monitoring Committee (IDMC) conducted a preliminary evaluation of the safety. If approved by the IDMC after the safety evaluation, the trial will proceed to the second stage. Before the result of the interim analysis are obtained, subjects receiving APL-1202 will continue to be given continuous administration if they have completed the 6-month visit (V4). After the interim analysis, if the safety of continuous administration is as expected, subjects receiving APL-1202 will continue to do the same, otherwise it will be adjusted to the administration of APL-1202 at every 3-month interval which is proven to be safe and tolerable.

• Second stage: After the interim analysis of the first stage, the subjects of the second stage will be enrolled, and the subjects were randomly assigned to receive APL-1202 single-agent oral treatment or intravesical instillation of Epirubicin hydrochloride at a ratio of 1:1. For treatment, according to the results of the interim analysis, if the safety of continuous administration reaches the expected level, subjects receiving APL-1202 will continue to do the same, otherwise it will be adjusted to the administration of APL-1202 at every 3-month interval which is proven to be safe and tolerable.

In this trial, the APL-1202 dosing regimen will continue until subjects exit the trial early for any reason, complete 24 months' treatment or the trial is terminated early.

Cystoscopy will be performed every 3 months in the enrolled subjects. If there is no recurrence in the enrolled subject during the treatment period (2 years after enrollment), cystoscopy will be performed every 6 months during the follow-up period until recurrence or the end of the clinical trial.

Safety assessment will be performed every 3 months during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all the following criteria:

* Must be informed of the investigational nature of this study and must provide written informed consent
* Age ≥18 years, male or female
* Non-muscle invasive transitional cell carcinoma of the bladder is histologically confirmed by Independent Pathology Review Committee (IPRC). Diagnosis and classification of intermediate-risk NMIBC is according to 2014 CUA Guideline of Diagnosis and Treatment of Urological Diseases in China:

Low-risk: Primary, solitary, TaGl (PUNLMP, low-grade urothelial carcinoma), <3cm, no CIS. (Note: the above conditions must be met at the same time as a low-risk NMIBC) Intermediate-risk: All tumours not defined in the two adjacent categories (between the category of low and high risk) High-risk: Any of the following: ① T1 tumour; ②G3(high-grade urothelial carcinoma) tumour;③carcinoma in situ (CIS); ④ Multiple, recurrent and large (> 3 cm) TaG1G2(low-grade urothelial carcinoma) tumours (all features must be present)

• No visible tumor after transurethral resection of bladder tumor (TURBT) on tumor lesion. Some requirements about Re-TURBT are as follows: It is recommended to conduct the secondary TURBT under following situations: incomplete first TURBT; no muscle tissue found in the first TURBT specimen, except Ta G1 (low grade) tumor and CIS only.

The secondary TURBT is recommended 2-6 weeks, but better at 4 weeks, after the first TURBT.

For subjects undergoing secondary TURBT, they will be enrolled after the second TURBT

* Subjects who never received intravesical instillation (including BCG or intravesical chemotherapy) prior to enrollment, except single, immediate, post-operative intravesical chemotherapy.
* Willing to provide pathological tissue specimen for assessment
* ECOG PS ≤ 1
* Patients, who have not received blood transfusion or colony-stimulating factor treatment within 14 days before the examination, must have normal organ and marrow function within 42 days of study entry (according to normal range in clinical site).

Absolute neutrophil count >1.5×109/L Platelets > 100 ×109/L Hemoglobin > 9.0 g/dL Alkaline phosphatase < 2.5 ULN GFR (Cockcroft-Gault formula calculated) ≥ 50 mL/min Total bilirubin, alanine aminotransferase or aspartate aminotransferase< 1.5 ULN INR <1.5, except for subjects receiving anticoagulation therapy

* Female should be either surgically sterilized or menopause or agree to use effective contraceptive measures during treatment. Women of reproductive age must have a negative result of pregnancy test during the screening period (pregnancy test will be not required if one of the following situations exists: the subject has undergone sterilization such as hysterectomy and/or bilateral oophorectomy, has no menstruation for 12 months and been diagnosed as menopause based on factors such as age). However, pregnancy tests are required for patients with bilateral fallopian tube ligation.
* Male subjects should be either surgically sterilized or agreed to use effective contraceptive measures. From signing the informed consent, subjects must take continuous measures until 3 months after the end of the treatment of trial. The definition of effective contraceptive measures will be based on the principal investigator(PI) or appointed delegate.
* Expected life expectancy is more than 48 months

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

* Low-risk: Primary, solitary, TaGl (PUNLMP, low-grade urothelial carcinoma), <3cm, no CIS. (PS: the above conditions must be met at the same time as a low-risk NMIBC)
* High-risk: Any of the following: ① T1 tumour; ②G3(high-grade urothelial carcinoma) tumour;③carcinoma in situ (CIS); ④ Multiple, recurrent and large (> 3 cm) TaG1G2(low-grade urothelial carcinoma) tumours (all features must be present)
* Tumors of T2 stage or more serious
* The histological types are mainly non-urothelial carcinomas such as squamous cell carcinoma and adenocarcinoma
* Urothelial carcinoma outside the bladder (renal pelvis, ureter or urethra)
* Received intravesical therapy in last TURBT/cystoscopy prior to treatment period, but not including immediate intravesical therapy once (the subjects who received the immediate intravesical therapy need to be recorded in e-CRF)
* Received surgery (not includes TURBT/cystoscopy), radiation therapy, or systemic therapy within 6 weeks before enrollment
* Malignancies within 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ' of the cervix
* Grade 3 (according to the NCI CTCAE 5.0) hemorrhage in any part of body within 6 weeks before starting the treatment of trial
* Any of the following within 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Hypertension that cannot be controlled by medications (systolic blood pressure≥140 mmHg and/or diastolic blood pressure≥90mmHg)
* Uncontrolled active infections before starting the treatment of trial, such as acute pneumonia, active hepatitis B, etc.
* Dysphagia or known drug absorption disorders
* Anuria
* One week prior to enrollment, having gross hematuria
* Active duodenal ulcers, ulcerative colitis and other gastrointestinal diseases or other conditions that the investigator may determine to cause gastrointestinal bleeding or perforation
* The risk of participation or administration may increase, judged by investigator, or other severe acute or chronic medical conditions may interfere with the interpretation and judgment of results
* or optic nerve disorders
* Subjects have optic nerve disorders and cataracts, or other related medical history
* Pregnancy or breastfeeding. Female patients with reproductive potential have a positive pregnancy test prior to enrollment
* Psychological or mental abnormality, subjects are estimated to have insufficient adherence to this clinical study
* Four weeks prior to enrollment, participate in other clinical trials
* Patients who had previously received anthracycline for systemic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 48 months
  Event-free survival (EFS) based on the assessment of pathological report from the Independent Pathology Review Committee (IPRC)

SECONDARY OUTCOMES:
Event-free survival (EFS) based on the assessment of pathological report from each site | Up to 48 months
  Event-free survival (EFS) based on the assessment of pathological report from each site
Overall survival (OS) | Up to 48 months
  Overall survival (OS)
Recurrence-free rate | Up to 48 months
  Recurrence-free rate at 12,18, and 24 months after enrollment
Progression-free rate | Up to 48 months
  Progression-free rate at 12,18, and 24 months after enrollment
Clinical benefit rates | Up to 48 months
  Clinical benefit rates at 12,18, 24 months after enrollment (clinical benefits are defined as the pathological improvement of the recurrence, no high-risk recurrence, progression-free recurrence, no radical therapy and no death)
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life Total Score | Up to 48 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall outcome
Change from Baseline in EORTC-QLQ-Non-muscle Invasive Bladder Cancer Module 24 (NMIBC24) Total Score | Up to 48 months
  The EORTC-QLQ-NMIBC24 is a 24-item questionnaire developed to supplement the EORTC QLQ-C30 in high-risk NMIBC patients. Each item is scored out of 4 total points (1=Not at All to 4=Very Much). All responses are transformed from 0 to 100, with a high score indicating more symptoms or problems. The change from baseline in EORTC-QLQ-NMIBC24 total score will be presented.

OTHER OUTCOMES:
Cystectomy-free survival (CFS) | Up to 48 months
  Cystectomy-free survival (CFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No